CLINICAL TRIAL: NCT00622115
Title: A Phase I, Pharmacokinetic and Tolerability Study of Intravenous Unfractionated Heparin After Subcutaneous Enoxaparin 1mg/kg Bid Repeated Administration in Healthy Subjects
Brief Title: Etude (Study) Phase I Enox - UnFractionated Heparin (UFH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Kazuki Otani/ Medical Project Manager, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENOXA_C_02537; 2007-000884-99
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Enoxaparin

ARMS (3):
- A (Experimental): 70 U/kg of UnFractionated Heparin (UFH) administered intravenously at 4 hours following the last injection of enoxaparin
  Interventions: Drug: Enoxaparin
- B (Experimental): 70 U/kg of UnFractionated Heparin (UFH) administered intravenously at 6 hours following the last injection of enoxaparin
  Interventions: Drug: Enoxaparin
- C (Experimental): 70 U/kg of UnFractionated Heparin (UFH) administered intravenously at 10 hours following the last injection of enoxaparin
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
Primary objective:

* to characterize the pharmacokinetic and the pharmacodynamic profile after intravenous bolus injection of unfractionated heparin (UFH) after repeated sc 100 IU anti-Xa/kg (corresponding to 1 mg/kg) twice a day during 2.5 days (every 12±2hrs) administrations of enoxaparin in Caucasian healthy subjects.

Secondary objective(s):

* to compare the pharmacokinetic and the pharmacodynamic profile between 3 different timing of administration of the UFH
* to assess the tolerability of the different anticoagulation protocols

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Male and female subjects, between 40 and 60 years of age
* Body weight between 50 kg and 90 kg if male and between 40 and 80 kg if female with Body Mass Index (BMI) between 18 and 29 kg/m2

Health Status:

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination)
* Subject with hypertension, hypo- or hyperthyroidism or dyslipidemia will be included if their concomitant pathology is well-controlled by treatment for at least one year
* Normal vital signs after 10 minutes resting in supine position:

  * 95 mmHg < systolic blood pressure (SBP) < 140 mmHg;
  * 45 mmHg < diastolic blood pressure (DBP) < 90 mmHg;
  * 40 bpm < heart rate < 100 bpm.
* Normal 12-lead electrocardiogram (ECG); 120 ms < PR < 220 ms, QRS < 120 ms, QTc ≤ 430 ms for male, 450 ms for female or not considered as clinically significant by the investigator
* Laboratory parameters within the normal range unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; hepatic enzymes (aspartate amino-transferase or AST, alanine amino-transferase or ALT) should be strictly below the upper laboratory norm.
* Platelets ≥ 150 000 / mm3
* Mean corpuscular volume (MCV) and gamma glutamyl-transferase (GGT) should be strictly in the normal range of the laboratory
* Activated partial thromboplastin time (aPTT) ratio should be comprised between 0.95 and 1.15
* Estimated Creatinine clearance by Cockroft formula should be higher than 50 mL/min
* Non smoker or smoking the equivalent or less than 5 cigarettes a day and able not to smoke during the study hospitalization
* Normal gynecological examination no longer than 12 months before inclusion.
* For female with childbearing potential using an effective contraception method (e.g. intra-uterine device, hormonal contraception, diaphragm and condom) except if postmenopausal for more than 12 months or sterilized for more than three months
* Subject with coagulation test and blood count (including platelets) within the physiological ranges)

Regulations:

* Having given written informed consent prior to any procedure related to the study
* Covered by Health Insurance System and/or in compliance with the recommendations of National Law in force relating to biomedical research
* Not under any administrative or legal supervision

Exclusion Criteria:

Medical history and clinical status:

* Contra-indication to anticoagulant therapy
* Subject with known increased bleeding time, hemophilia, thrombocytopenia, and/or history of any vascular purpura
* Subject with detectable antibody against heparin in the blood
* Any history or presence of clinically relevant cardiovascular, gynecologic (for women), pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, ocular or infectious disease that is capable of altering the absorption, metabolism, or elimination of drugs, or of constituting a risk factor when taking the study medication; any acute infectious disease or signs of acute illness; except subject with hypertension, hypo- or hyperthyroidism or dyslipidemia if well-controlled by treatment for at least one year.
* Subject with diabetes or other cardiovascular or metabolic disease
* Subject with INR > 1.5
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month)
* Blood donation or blood loss within one month before administration
* Symptomatic hypotension whatever the decrease in blood pressure or asymptomatic postural hypotension defined by a decrease in SBP equal to or greater than 20 mmHg within three minutes when changing from the supine to the standing position
* Presence or history of drug allergy, or allergic disease diagnosed and treated by a physician
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams/day)
* Smoking more than 5 cigarettes or equivalent/day, or unable to stop smoking during the study
* Excessive consumption of beverages with xanthine bases (> 4 cups or glasses/day)
* Pregnancy (defined as positive beta-HCG plasma test that can not be explicated by menopauses), breast-feeding for female, any history or presence of clinically relevant gynecologic disease

Interfering substance:

* Any medication (including St John's Wort) within 14 days before administration, or within 5 times the elimination half-life of that drug, except for hormonal contraception or replacement therapy, and allowed therapy for stable pathology
* Anti-inflammatory treatments and anti-aggregant treatments are strictly forbidden during the whole study period

General conditions:

* Subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development
* Subject in exclusion period of a previous study according to applicable regulations
* Subject who cannot be contacted in case of emergency
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff thereof, directly involved in the conduct of the protocol or any other protocol of the Investigating Center
* Subject is an employee of the Investigating Center

Biological status:

* Positive reaction to any of the following tests: HBs antigen, anti-HCV antibodies, anti-HIV1 antibodies, anti-HIV2 antibodies, anti-LMWH antibodies
* Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids)
* Positive alcohol breath or plasma test

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Concentration-time profiles of anti-Xa and anti-IIa levels | At baseline (Day 2) after the morning enoxaparin injection and at day 3 from pre-dose of enoxaparin and lasting until 14 hours after the enoxaparin injection.

SECONDARY OUTCOMES:
Effect-time profiles of ACT, TGTppp and TGTprp | At baseline (Day 2) after the morning enoxaparin sc injection and at day 3 from pre-dose of enoxaparin and lasting until 14 hours after the enoxaparin injection.
PFA100 levels measured | At pre-dose, 4h and 14h post dose of enoxaparin
Documentation of adverse event, physical examination, clinical laboratory safety, vital signs and ECG recording at prespecified time-points. | during the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Otani, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France

REFERENCES:
- [Background] Drouet L, Bal dit Sollier C, Martin J. Adding intravenous unfractionated heparin to standard enoxaparin causes excessive anticoagulation not detected by activated clotting time: results of the STACK-on to ENOXaparin (STACKENOX) study. Am Heart J. 2009 Aug;158(2):177-84. doi: 10.1016/j.ahj.2009.05.022. PMID 19619692